CLINICAL TRIAL: NCT01118702
Title: A Randomized, Open-label, Single-dose, Three-way Crossover Study to Determine the Relative Pharmacokinetic Profile of Oral Doses of CONCERTA Tablets, Ritalin-SR Tablets and Novo-Methylphenidate ER-CTablets Under Fasted Condition in Healthy Subjects
Brief Title: A Study to Explore Plasma Levels of CONCERTA, Ritalin-SR and Novo-Methylphenidate ER-C in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR017179; CR017179 (Other: Janssen-Ortho, Canada)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetic; Methylphenidate; Novo-methylphenidate ER-C; Ritalin-SR; CONCERTA; Plasma profile
MeSH Terms: interventions — Methylphenidate

ARMS (3):
- 001 (Active Comparator): Concerta one 54mg tablet once
  Interventions: Drug: Concerta
- 002 (Active Comparator): Ritalin-SR 3-20mg tablets once
  Interventions: Drug: Ritalin-SR
- 003 (Active Comparator): Novo-Methylphenidate ER-C one 54mg tablet once
  Interventions: Drug: Novo-Methylphenidate ER-C

INTERVENTIONS:
Drug: Ritalin-SR — 3-20mg tablets, once
  Arms: 002
Drug: Concerta — one 54mg tablet, once
  Arms: 001
Drug: Novo-Methylphenidate ER-C — one 54mg tablet, once
  Arms: 003

SUMMARY:
This is a study of blood plasma levels of methylphenidate in healthy volunteers over a 24 hour period after they take this medication.

DETAILED DESCRIPTION:
The purpose of this study is to measure the blood plasma concentrations of methylphenidate in healthy volunteers for 24 hours after they take three different long acting methylphenidate products. This is a single-centre, randomized (subjects will be assigned a treatment sequence based on chance), open-label (all people involved know the identity of the intervention), single-dose, three-way crossover study (participants may receive different interventions sequentially during the trial) in 30 healthy adult volunteers. Study drug will be taken by mouth with 240mL of room temperature noncarbonated water. Blood sampling will be done via indwelling catheter at pre dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 11, 12, 14, 16, 20 and 24 hours post dose. An indwelling venous catheter is put in place for the 24 hour period to minimize the discomfort of frequent blood sampling. Each patient will receive one dose of each treatment under study in a specific sequence and at specified timepoints. The treatments are: one 54mg Concerta tablet, one 54 mg Novo-methylphenidate ER-C tablet, and 3x20mg Ritalin-SR tablets. The methylphenidate plasma concentrations observed during the 24 hour post-dose time period will be compared for each volunteer and across all volunteers. Adverse events will be monitored from the time the informed consent is signed until the patient completes the last study-related procedure. The investigator must follow all adverse events reported to the investigator to satisfactory resolution or until reaching a clinically stable endpoint. Vital signs will be taken at study entry and before each dose - as well as at specific timepoints over the 24 hour sample period. Clinical labs and EKG will be done at screening and at each 24 hour timepoint.

The official study title is as follows: A Randomized, Open-label, Single-dose, Three-way Crossover Study to Determine the Relative Pharmacokinetic Profile of Oral Doses of CONCERTA Tablets, Ritalin-SR Tablets and Novo-Methylphenidate ER-C Tablets Under Fasted Condition in Healthy Subjects. Methylphenidate is indicated for the treatment of attention deficient hyperactivity disorder in adults, adolescents and children. Each volunteer will receive one 54-mg CONCERTA tablet(once), one 54-mg Novo-Methylphenidate ER-C tablet (once) and three 20mg Ritalin-SR tablets (once) at specified time points in the study. Tablets will be administered as a single oral dose under fasted (minimum 10 hour fast) conditions. Study drug will be administered orally with 240 mL of room temperature noncarbonated water.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer will be assessed against all protocol specified criteria at investigator site: If a female, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives for at least 3 months, contraceptive injections, intrauterine device, contraceptive patch, male partner sterilization) before entry, throughout the study, and 1 week after the completion of the study
* if female, must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening and on Day -1 of each treatment period
* Body mass index (weight [kg]/height [m2]) between 18 and 30 kg/m2 (inclusive)
* Body weight not less than 50 kg
* Blood pressure (after the patient is sitting for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and 50 and 90 mmHg diastolic, inclusive

Exclusion Criteria:

* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, birth control (prescription oral contraceptives, contraceptive injections, intrauterine device, contraceptive patch), and hormonal replacement therapy within 14 days before the first dose of the study drug
* Current, history or a reason to believe a subject has a history of drug or alcohol abuse/dependence according to DSM-IV
* Positive test for drugs of abuse
* Known allergy to the study drug or any of the ingredients in the study drug tablets
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half life, whichever is longer, before the first dose of the study drug - a drug's half life is the time that it takes the body to excrete 50% of the drug
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)
* If a female, breast-feeding or planning to become pregnant during the study or within 60 days of last study drug
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies administration
* History of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or patient's verbal report
* May not consume food or beverages containing alcohol, grapefruit juice, Seville oranges, or quinine (e.g., tonic water) from 24 hours (72 hours in the case of grapefruit juice and Seville oranges) before each PK sample collection day, until after the last PK sample is collected in each period
* Must refrain from the use of any methylxanthine-containing products, (e.g., chocolate bars or beverages, coffee, teas, or colas) from 48 hours before administration of study drug and during confinement, and when caffeine is allowed, must avoid excessive use of caffeine (i.e., no more than approximately 500 mg/day, as contained in 5 cups of tea or coffee or 8 cans of cola), during the entire study (from screening to end of study)
* May not consume food containing poppy seeds during the study
* Must refrain from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch) throughout the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this exploratory study is to characterize the plasma concentrations of of methylphenidate from Concerta®, Ritalin-SR® and Novo-Methylphenidate ER-C ® tablets in healthy adult volunteers under fasting conditions. | Plasma samples will be taken via in-dwelling catheter predose, and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 11, 12, 14, 16, 20 and 24 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Derived] Shram MJ, Quinn AM, Chen N, Faulknor J, Luong D, Sellers EM, Endrenyi L. Differences in the in vitro and in vivo pharmacokinetic profiles of once-daily modified-release methylphenidate formulations in Canada: examination of current bioequivalence criteria. Clin Ther. 2012 May;34(5):1170-81. doi: 10.1016/j.clinthera.2012.02.010. Epub 2012 Apr 17. PMID 22512898
- See also: A Randomized, Open-label, Single-dose, Three-way Crossover Study to Determine the Relative Pharmacokinetic Profile of Oral Doses of CONCERTA® Tablets, Ritalin-SR® Tablets and Novo-Methylphenidate ER-C® Tablets under Fasted Condition in Healthy Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=374&filename=CR017179_CSR.pdf